CLINICAL TRIAL: NCT01304602
Title: A Phase I Trial of Irinotecan and BKM120 in Previously Treated Advanced Colorectal Cancer
Brief Title: A Trial of Irinotecan and BKM120 in Previously Treated Advanced Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12480
Record Dates: First submitted 2011-02-18; First posted 2011-02-25 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; BKM120; irinotecan
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; NVP-BKM120

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Irinotecan + BKM120 (Experimental): Irinotecan + BKM120 at the assigned cohort dose level.
  Interventions: Drug: Irinotecan; Drug: BKM120

INTERVENTIONS:
Drug: Irinotecan — IV over 90 minutes on day 1 of each cycle (every 2 weeks) at the cohort assigned dose level
  Other Names: Camptostar
Drug: BKM120 — BKM120, oral, daily starting with cycle 1/day 2 at the cohort defined dose level

SUMMARY:
This phase I trial will use the combination of irinotecan and BKM120 in patients with advanced colorectal cancer who have failed on or have become intolerant of at least one line of therapy for advanced colorectal cancer and who are candidates for irinotecan therapy.

DETAILED DESCRIPTION:
Although survival of patients with advanced colorectal cancer has improved in the last two decades, the overwhelming majority of these patients will still succumb from this disease. It is the third most commonly diagnosed malignancy in the United States. We have witnessed significant leaps in understanding colorectal cancer carcinogenesis as well as in identification of a number of prognostic and predictive factors associated with this malignancy. With the use of combination chemotherapy and the addition of targeted agents, the median survival of patients with advanced colorectal cancer has improved from 4-6 months with supportive care to over 2 years.

Molecularly directed therapy for cancer holds promise to a more personalized approach to treating cancer. Increase understanding of tumorigenesis has resulted in the identification of promising targets of therapy for more strategic approach to treatment of this malignancy. However, even with the development of molecularly directed treatment, the therapy for advanced colorectal cancer remains to be primarily palliative in nature to majority of patients. There is definite need for a more effective therapy, agents with more acceptable toxicity profiles, and drugs that could be administered without significant demand on time and activity for individual patients receiving these drugs.

This is a phase I trial of the combination of irinotecan and BKM120 in patients with advanced colorectal cancer who have failed on or have become intolerant of at least one line of therapy for advanced colorectal cancer and who are candidates for irinotecan therapy. This study will attempt to estimate the Maximum Tolerated Dose of the combination of irinotecan and BKM120.

ELIGIBILITY:
Inclusion Criteria

* Histologically or cytologically confirmed metastatic or unresectable adenocarcinoma of the colon or rectum with measurable disease (patients who have become resistant or intolerant of at least one-line of chemotherapy regimen are eligible)
* Patients who had had previous treatment with Irinotecan and who have definite progression on Irinotecan are eligible provided they are not a candidate for other therapeutic treatment options. Definitive progression is defined as progression of disease while on Irinotecan or within 4 weeks of discontinuing Irinotecan.
* ≥ 18 years old
* ECOG performance status ≤ 2 (Karnofsky > 60%)
* ANC ≥ 1.5 x 109/L, Platelets ≥ 100 x 109/L, Hb >9 g/dL
* Serum bilirubin within normal range (or < 1.5 x IULN if liver metastases present; or total bilirubin ≤ 3.0 x IULN with direct bilirubin within normal range in patients with well documented Gilbert Syndrome)
* AST (SGOT) or ALT (SGPT) within normal range (or ≤ 3.0 x upper limit of normal if liver metastases present)
* adequate renal function as evidenced by creatinine ≤ 1.5 x IULN or creatinine clearance ≥ 50 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal.
* serum calcium (corrected for serum albumin) within normal limits. Biphosphonate use for malignant hypercalcemia control is not allowed.
* Serum magnesium ≥ the institutional lower limit of normal (ILLN) and potassium within institutional normal limits.
* serum lipase ≤ IULN; serum amylase ≤ IULN; fasting plasma glucose ≤ 120 mg/dL (6.7 mmol/L)
* females of child-bearing potential must have negative serum pregnancy test within 72 hours prior to treatment. Cannot be pregnant or nursing.
* Males and females must agree to use effective contraceptive method.
* INR ≤ 2 Exclusion Criteria
* Previous treatment with chemotherapy, biologic therapy, or wide field radiotherapy < 4 weeks or limited field radiation for palliation < 2 weeks prior to starting study drug; must have recovered from side effects of such therapy
* Known hypersensitivity to BKM120 or to its excipients or to irinotecan
* Untreated brain metastases. Patients with metastatic CNS tumors may participate in this trial, if the patient is > 4 weeks from therapy completion, is clinically stable and is not receiving corticosteroid therapy
* Known polymorphism in UGTAIA or Gilbert's syndrome
* Acute or chronic liver, renal disease or pancreatitis
* Medically documented history or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, history of suicidal attempt or ideation, or homicidal ideation; ≥ CTCAE grade 3 anxiety; meets cutoff score of ≥ 10 in the PHQ-9 or cut-off of ≥ 15 in GAD-7 mood scale, respectively, or selects positive response of "1, 2, or 3" to question number 9 regarding potential for suicidal thoughts in the PHQ-9 (independent of the total score of the PHQ-9)
* Clinically significant heart disease including: Left ventricular ejection fraction (LVEF) <50% as determined by echocardiogram; ventricular arrhythmias except for benign premature ventricular contractions; supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication; conduction abnormality requiring a pacemaker; valvular disease with documented compromised cardiac function; symptomatic pericarditis; QTc > 480 msec on screening ECG (using QTcF formula; angina pectoris that requires use of anti-anginal medication
* History of cardiac dysfunction including: acute myocardial infarction ≤ 6 months, documented by persistent elevated cardiac enzymes or persistent regional wall abnormalities on assessment of LVEF function; history of documented congestive heart failure (NYHA Class III or IV; document cardiomyopathy
* Other concurrent severe and/or uncontrolled concomitant medical conditions
* Significant symptomatic deterioration of lung function. If clinically indicated, pulmonary function tests including measures of predicted lung volumes, DLco, O2 saturation at rest on room air should be considered to exclude pneumonitis or pulmonary infiltrates
* Clinical manifestation of diabetes mellitus or steroid-induced diabetes mellitus
* Impairment of GI function or disease that may significantly alter the absorption of BKM120; diarrhea ≥ grade 2
* Major surgery ≤ 4 weeks prior to starting study drug
* Prior treatment with a P13K inhibitor; any hematopoietic colony-stimulating growth factors ≤ 2 weeks prior to starting study drug; corticosteroids ≤ 2 weeks prior to starting study drug; chemotherapy or targeted anticancer therapy ≤4 weeks (6 weeks for nitrosourea, antibodies or mitomycin-C) prior to starting study drug; small molecule therapeutics (excluding monoclonal antibodies) ≤5 effective half-lives prior to starting study drug
* Currently receiving medication that has the potential to prolong the QT interval or inducing Torsades de Pointes
* chronic treatment with steroids or another immunosuppressive agent. Note: Topical applications (eg rash), inhaled sprays (eg obstructive airways diseases), eye drops or local injections (eg intra-articular) are allowed. Patients with previously treated brain metastases, who are on stable low dose corticosteroids treatment (eg dexamethasone 2 mg/day, prednisolone 10 mg/day) for at least 14 days before start of study treatment are eligible.
* therapeutic doses of warfarin sodium or any other coumadin-derivative anticoagulant.
* any medications or substances that are inhibitors or inducers of specific CYP450 enzyme(s).
* any other study agents
* Patients who have taken herbal medications and certain fruits within 7 days prior to starting study drug. Herbal medications include, but are not limited to St. John's wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng. Fruits include the CYP3A inhibitors Seville oranges, grapefruit, pummelos, or exotic citrus fruits.
* Patients who have received wide field radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Women who are pregnant or breast feeding; adults of reproductive potential not using an effective method of birth control.
* Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (eg age appropriate, history of vasomotor symptoms) or 6 months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL and estradiol < 20 pg/mL or have had surgical bilateral oophorectomy (with or without hysterectomy) at least 6 weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, must use highly effective contraception during treatment for 8 days after stopping treatment and for additional 12 weeks after study drug discontinuation. Highly effective contraception is defined as: true abstinence: Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception. Sterilization: have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least 6 weeks ago. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
* Male partner sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). For female subjects on the study, the vasectomised male partner should be the sole partner for that patient.
* Use of a combination of any two of the following (a+b): Placement of an intrauterine device (IUD) or intrauterine system (IUS); Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository; Oral contraception, injected or implanted hormonal methods are not allowed as BKM120 potentially decreases the effectiveness of hormonal contraceptives.
* Fertile males must use condom during treatment, for 8 days after stopping treatment and for additional 12 weeks after study drug discontinuation and should not father a child in this period.
* Known diagnosis of human immunodeficiency virus (HIV) infection
* History of another malignancy within 3 years, except cured basal cell skin carcinoma or excised cervical carcinoma in situ
* Previous treatment with Irinotecan who have definite progression on Irinotecan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-02; Primary Completion 2014-04 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 28 days
  The maximum tolerated dose will be defined as the dose level prior to the dose level in which dose-escalation was stopped based on dose-limiting toxicities (DLTs). DLTs are based on specific adverse events specified in the study protocol. DLTs will be assessed during the first two cycles of treatment (28 days total).

SECONDARY OUTCOMES:
area under the plasma concentration versus time curve (AUC) of irinotecan | up to 25.5 hours post dose of irinotecan
  Blood samples will be collected at cycle 1/day 1 and cycle 2/day 1 to determine the AUC of irinotecan in the presence and absence of BKM120.
Change in tumor size | baseline, and every 8 weeks
  Disease will be assessed at baseline and then every four cycles (8 weeks) by CT or MRI. Response will be assessed following RECIST criteria. Patients will be categorized as complete response, partial response, progressive disease, stable disease, or unknown.
Peak Plasma Concentration (Cmax) of irinotecan | up to 25.5 hours post-dose of irinotecan
  Blood samples will be collected at cycle 1/day 1 and cycle 2/day 1 to determine the AUC of irinotecan in the presence and absence of BKM120.
biological half-life of irinotecan | up to 25.5 hours post dose of irinotecan
  Blood samples will be collected at cycle 1/day 1 and cycle 2/day 1 to determine the AUC of irinotecan in the presence and absence of BKM120.
Peak Plasma Concentration (Cmax) of BKM120 | up to 25.5 hours post-dose of irinotecan
  The Cmax of BKM120 will be measured at Cycle 2/Day 1 for pharmacokinetic characterization of BKM120.
area under the plasma concentration versus time curve (AUC) of BKM120 | up to 25.5 hours post dose of irinotecan
  The AUC of BKM120 will be measured at Cycle 2/Day 1 for pharmacokinetic characterization of BKM120.
Biological half life of BKM120 | up to 25.5 hours post dose of irinotecan
  The biological half life of BKM120 will be measured at Cycle 2/Day 1 for pharmacokinetic characterization of BKM120.

CONTACTS AND LOCATIONS:
Overall Officials: Joaquina Baranda, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Cancer Center, Kansas City, Kansas, United States